CLINICAL TRIAL: NCT05872555
Title: Side Effects of Psychiatric Medications - a Nested Case Control Cohort Historical Prospective Study
Status: Active, not recruiting | Type: Observational
Sponsor: Mark Weiser, MD, Principal Investigator (Other Government)
Responsible Party: Sponsor-Investigator, Mark Weiser, MD, Principal Investigator, Head of Psychiatry, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Other Study IDs: 0277-23-SMC
Record Dates: First submitted 2023-05-09; First posted 2023-05-24 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Psychotic Disorders
Keywords: Antipsychotics; Side effects; Metabolic
MeSH Terms: conditions — Psychotic Disorders | interventions — Antipsychotic Agents; Benzodiazepines; Antidepressive Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with psychiatric diagnosis/prescribed psychiatric medications: 1. Diagnosed with schizophrenia/schizoaffective disorder/bipolar disorder/depression/dementia/diagnosed with other psychiatric disorders, or not diagnoses with any disorder, and registered in the Clalit database.
  2. First exposure to antipsychotics/antidepressants/benzodiazepines/mood stabilizers above the age of 16 years, regardless of the presence of having a psychiatric diagnosis. We will include patients treated with these medications also if they do not have a psychiatric diagnosis.
  3. Prescription of these psychiatric medications between 2001-2024
  Interventions: Drug: Psychiatric Drugs
- Control individuals: 1. The control groups will differ according to the analysis performed, and will be clearly described in the publication.
  2. Depending on the analysis, will not include person prescribed antipsychotics, antidepressants, benzodiazepines, mood stabilizers.
  3. Matched for age, sex and socio-economic status and other potential confounders, depending on the disease studied.

INTERVENTIONS:
Drug: Psychiatric Drugs — Receiving any Antipsychotic, Benzodiazepine, antidepressant, mood stabilizer
  Other Names: Antipsychotics, Benzodiazepines, antidepressants, mood stabilizers
  Groups: Patients with psychiatric diagnosis/prescribed psychiatric medications

SUMMARY:
The study is designed to fill in the gaps in current knowledge by providing a more inclusive and comprehensive understanding of the potential associations between different psychiatric medications, including antipsychotics (APs), Antidepressants, Benzodiazepines and mood stabilizers, and negative outcomes, as previous research has often been limited to data from clinical trials.

The primary objectives of the study include assessing the association between different psychiatric medications and long-term major negative medical conditions and events. Additionally, the study aims to assess the association between different psychiatric medications and long-term negative metabolic events such as diabetes, obesity, hypertension and hypercholesterolemia.

This study aims to investigate the potential long-term negative effects of different psychiatric medications on patients with schizophrenia, schizoaffective disorder, depression, bipolar disorder and dementia, patients with other diagnoses, as well as patients receiving different psychiatric medications who do not have a psychiatric diagnosis. The study will be done using data from the Clalit Health Services (CHS) database, which is the largest provider of health insurance in Israel, serving approximately 55% of the population. This database provides access to all diagnoses and blood tests for the duration of the study, which allows for accurate tracking of patient outcomes over time.

Inclusion criteria include being diagnosed with schizophrenia/schizoaffective disorder/bipolar disorder/depression, dementia, other psychiatric diagnoses, and/or patients receiving these medications who do not have a psychiatric diagnosis, and use psychiatric medications, including antipsychotics/antidepressants/mood stabilizers/benzodiazepines as registered in the Clalit database. having first prescription of psychiatric medication between 2001 and 2024. The study will look at those patients included and will follow them using the CHS database to assess these different medical and or metabolic side-effects and the appearance of major negative and major metabolic events, as well as abnormal metabolic measurements.

DETAILED DESCRIPTION:
The study is designed to fill in the gaps in current knowledge by providing a more inclusive and comprehensive understanding of the potential associations between different psychiatric medications, including antipsychotics (APs), Antidepressants, Benzodiazepines and mood stabilizers, and negative outcomes, as previous research has often been limited to data from clinical trials.

The primary objectives of the study include assessing the association between different psychiatric medications and long-term major negative events such as cancer, osteoporosis, hip fracture, acute myocardial infarction, stroke, tardive dyskinesia, chronic obstructive pulmonary disease, chronic kidney failure and dialysis. Additionally, the study aims to assess the association between different psychiatric medications and long-term negative metabolic events such as diabetes, obesity, hypertension and hypercholesterolemia The study also aims to assess the association between different psychiatric medications and long-term negative metabolic measurements such as increased body mass index, cholesterol levels, triglyceride levels, Hemoglobin A1C levels and glucose levels, hyperprolactinemia, as well as low eGFR.

This study aims to investigate the potential long-term negative effects of different psychiatric medications on patients with schizophrenia, schizoaffective disorder, depression, bipolar disorder and dementia, patients with other diagnoses, as well as patients receiving different psychiatric medications who do not have a psychiatric diagnosis. The study will be done using data from the Clalit Health Services (CHS) database, which is the largest provider of health insurance in Israel, serving approximately 55% of the population. This database provides access to all diagnoses and blood tests for the duration of the study, which allows for accurate tracking of patient outcomes over time.

Inclusion criteria include being diagnosed with schizophrenia/schizoaffective disorder/bipolar disorder/depression, dementia, other psychiatric diagnoses, and/or patients receiving these medications who do not have a psychiatric diagnosis, and use psychiatric medications, including antipsychotics/antidepressants/mood stabilizers/benzodiazepines as registered in the Clalit database. having first prescription of psychiatric medication between 2001 and 2024. The study will look at those patients included and will follow them using the CHS database to assess these different medical and or metabolic side-effects and the appearance of major negative and major metabolic events, as well as abnormal metabolic measurements.

The preliminary analysis of the study used a sample of 22,777 patients diagnosed with schizophrenia or schizoaffective disorder between the years 2001-2021 in the Clalit dataset. This sample was used to assess whether patients who received at any time clozapine, olanzapine, and quetiapine had a higher risk of major negative and metabolic events. The analysis found that patients who received these medications were at a higher risk of developing metabolic outcomes and most major negative events. Based on these findings, the study aims to have a sample size large enough to detect these associations and allow for meaningful conclusions to be drawn from the data.

ELIGIBILITY:
Inclusion Criteria:

Study Group:

1. Diagnosed with schizophrenia/schizoaffective disorder/bipolar disorder/depression/dementia/diagnosed with other psychiatric disorders, or not diagnoses with any disorder, and registered in the Clalit database.
2. First exposure to antipsychotics/antidepressants/benzodiazepines/mood stabilizers above the age of 16 years, regardless of the presence of having a psychiatric diagnosis. We will include patients treated with these medications also if they do not have a psychiatric diagnosis.
3. Prescription of these psychiatric medications between 2001-2024

Control Group:

1. The control groups will differ according to the analysis performed, and will be clearly described in the publication.
2. Depending on the analysis, will not include person prescribed antipsychotics, antidepressants, benzodiazepines, mood stabilizers.
3. Matched for age, sex and socio-economic status and other potential confounders, depending on the disease studied.

Exclusion Criteria:

* Individuals not meeting the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria for patients include being diagnosed with schizophrenia/schizoaffective disorder/bipolar disorder/depression/other psychiatric diagnoses, and will also include patients receiving these medications who do not have a psychiatric diagnosis. Using psychiatric medications including antipsychotics/antidepressants/mood stabilizers/benzodiazepines as registered in the Clalit database. The study will look at those patients included and will follow them using the CHS database to assess different medical side-effects and the appearance of major negative and major metabolic events, as well as abnormal metabolic measurements.
  Psychiatric diagnoses by ICD 10 are included if assigned by a psychiatrist or registered following hospital discharge. The validity of these diagnoses has been verified in previous studies (Bieber et al., 2013).
Sampling Method: Non-Probability Sample
Enrollment: 22777 (Estimated)
Dates: Start 2023-03-26 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Long-term major negative events | During follow-up from 2000 to 2021
  Report in national database of cancer, heart disease (heart failure, MI), lung disease (COPD), Tardive dyskinesia, Neurological conditions (CVA, TIA, Epilepsy), , Osteoporosis, hip fracture, chronic kidney disease and dialysis. The database includes a list of reported diseases and major health events, with a score of 0 for no report and a score of 1 for diagnosis of disease.
Long-term metabolic events | During follow-up from 2000 to 2021
  Diagnosis of Diabetes, Obesity, Hypercholesterolemia, Hypertension. A diagnosis will be considered positive if it appears for at least two years. A composite score will be defined as the appearance of a diagnosis of one or more of the following: diabetes, obesity, hypertension, hypercholesterolemia and hypertriglyceridemia.
Long-term metabolic measurements- BMI | During follow-up from 2000 to 2021
  BMI report- using metric units (weight in km/square of height in meters)
Long-term metabolic measurements- Cholesterol levels | During follow-up from 2000 to 2021
  Report of cholesterol levels measured in millimoles per liter (mmol/L)
Long-term metabolic measurements- Triglycerides levels | During follow-up from 2000 to 2021
  Report of triglyceride levels measured in millimoles per liter (mmol/L)
Long-term metabolic measurements- HbA1C levels | During follow-up from 2000 to 2021
  Report of glycated hemoglobin (HbA1C) levels measured in millimoles per moles (mmol/mol)
Long-term metabolic measurements- glucose levels | During follow-up from 2000 to 2021
  Report of glucose levels measured in millimoles per liter (mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Psychiatry Department, Ramat Gan, Israel